CLINICAL TRIAL: NCT01326468
Title: A Pilot Study of Chemoradiotherapy Plus Temsirolimus (Torisel) for Advanced Head and Neck Cancer
Brief Title: Torisel in Addition to Standard Chemotherapy With Radiation for Advanced Head and Neck Cancer
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: funding
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10D.133; 2009-44 (Other: CCRRC); JT 1537 (Other: JeffTrial Number)
Record Dates: First submitted 2011-03-29; First posted 2011-03-30 (Estimated); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Head and Neck Cancer
Keywords: head and neck cancer; temsirolimus; cetuximab; cisplatin; radiation therapy
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — temsirolimus; Cetuximab; Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A - Temsirolimus with Cisplatin (Experimental): Temsirolimus with cisplatin, Erbitux and radiation therapy
  Interventions: Drug: Temsirolimus; Drug: Cetuximab; Drug: Cisplatin; Device: Radiation Therapy
- Cohort B - Temsirolimus (Experimental): Temsirolimus with Erbitux and radiation therapy
  Interventions: Drug: Temsirolimus; Drug: Cetuximab; Device: Radiation Therapy

INTERVENTIONS:
Drug: Temsirolimus — All patients will receive temsirolimus. The dose of temsirolimus in this study will range from 15-25 mg depending on the dose level. Temsirolimus will be infused over a 30-60 minute period once a week for the duration of radiation therapy.
  Other Names: Torisel; CCI-779
Drug: Cetuximab — All patients will receive cetuximab. An initial loading dose of cetuximab 400 mg/m2, intravenously over 120 minutes at least 4 days before radiation therapy but no more than 7 days before the start of radiation therapy.
  Thereafter, cetuximab will be infused at 250 mg/m2 dose over 60 minutes weekly for the duration of radiation therapy.
  Other Names: IMC-C225; Erbitux
Drug: Cisplatin — All patients in Cohort A will receive cisplatin. The dose will be 20 mg/m2 or 30 mg/m2 depending upon the dose level.
  Other Names: cisplatinum; cis-diamminedichloroplatinum(II); CDDP; Platinol; Platinol-AQ
  Arms: Cohort A - Temsirolimus with Cisplatin
Device: Radiation Therapy — Patients will be treated on a linear accelerator fitted with multi-leaf collimators with 1.6-2.3 Gy fractions delivered daily 5 days per week over 4-7 weeks to a cumulative dose of 66 Gy. A variance of +/- 10% in this nominal prescription dose is allowable and will depend on the extent of residual disease, at the discretion of the attending radiation oncologist.
  Other Names: IMRT; RT; radiation oncology; radiotherapy; XRT

SUMMARY:
Patients with advanced head and neck cancer is at high risk of recurrence at the primary site or in the neck. Part of normal treatment is to treat such patients with chemotherapy and radiation. The chemotherapy can include Erbitux. The purpose of this study is to treat such patients with an additional agent, Torisel. This study tests the doses of Torisel that can be safely administered together with radiation and chemotherapy.

DETAILED DESCRIPTION:
Approximately 30,000 new cases of local-regionally advanced head and neck carcinoma (HNC) and head and neck squamous cell carcinoma (HNSCC) are diagnosed each year for which surgery is either insufficient, non-curative or not feasible. For these patients, radiation therapy is the mainstay of treatment often with the use of concurrent chemotherapy and/or concurrent cetuximab therapy. Radiation therapy is also commonly employed in the post-operative setting for patients with high risk features predisposing to recurrent disease. Although progress has been made, the prominent pattern of failure among these aggressively treated patients remains loco-regional failure.

The epidermal growth factor receptor (EGFR), a member of the ErbB family of receptor tyrosine kinases, is abnormally activated in nearly all epithelial cancers, including HNC. Nearly all HNC expressing high levels of EGFR have been associated with poor outcomes. Radiation therapy can lead to increased expression of EGFR in cancer cells, and blockade of EGFR signaling has been shown to sensitize cells to ionizing radiation. The use of monoclonal antibodies directed against EGFR has a rich pre-clinical record. However, it was not until the publication of the Bonner trial that combined radiotherapy plus anti-EGFR therapy was shown to be successful in the clinic to treat HNSCC. This study showed that the addition of single agent cetuximab 250 mg/m2 given weekly with concurrent radiation therapy improved median overall survival from 29 to 49 months. Furthermore, progression-free survival was improved from 12 to 17.1 months. In addition, patients were able to tolerate the regimen with no difference in rates of mucositis. Other toxicities were also similar to radiotherapy alone, with the exceptions of a small risk of infusion reactions, and the common - but non-dose limiting - occurrence of an acneiform rash.

Temsirolimus is a specific inhibitor of the mammalian target of rapamycin (mTOR), an enzyme that regulates cell growth and proliferation. Temsirolimus prevents progression from the G1 phase to the S phase of the cell cycle through inhibition of mTOR, which is a novel mechanism of action for an anticancer drug. This is also important for concurrent treatment with radiation, since S-phase represents the most radiation resistant phase of the cell cycle.

Temsirolimus is a structural analog of sirolimus (rapamycin) that has been formulated for IV or oral administration for the treatment of various malignancies. Sirolimus was shown to have potent immunosuppressive as well as antifungal and antitumor properties. Its mechanism of action results in part from binding to an intracellular cytoplasmic protein, FK506 (tacrolimus) binding protein (FKBP)-12. The complex of sirolimus bound to FKBP-12 blocks the activity of mTOR.

Cetuximab is an important agent in the treatment of HNSCC; however its success may be limited by downstream signaling molecules which may up-regulate and cause the malignant phenotype to persist. MET proto-oncogene amplification has been hypothesized to lead to EGFR-independent activation of the PI3K-Akt-mTOR pathway through activation of HER3-dependent signaling. We hypothesize that attacking HNC at two key points in the cellular proliferation and survival system will maximize HNC cell killing and irradicate subpopulations of cells which may be able to bypass the EGFR inhibition with independent activation of the PI3K-Akt-mTOR pathway. The concomitant use of cetuximab and temsirolimus permits active inhibition of both EGF, and the VEGF pathway related with angiogenesis, with synergistic responses as seen in experimental models.

Although patients who have pre-existing renal or functional conditions - preventing the administration of cisplatin - receive cetuximab concurrently with radiation as standard of care, there is a clear phenomenon of the development of EGFR inhibitor resistance. Therefore, the ability to target one of the escape pathways of EGFR inhibitor resistance via blockade of the PI3K pathway, possibly in the synergistic manner, provides an important and novel method for achieving high rates of complete and durable response to treatment in patients who are unable to tolerate traditional chemotherapeutic agents.

In most patients who do not have pre-existing renal or functional conditions, cisplatin is considered the standard of care. However, given the relatively poor rates of disease free survival with platinum and radiation combinations, the Radiation Therapy Oncology Group (RTOG) 0522 phase III trial of a combination of accelerated radiation therapy with cisplatin and cetuximab was completed to accrual in March 2009. The results of that trial are still pending, although the fact that it closed to accrual indicates that it was a tolerable regimen.

In patients who can receive cisplatin, they will receive temsirolimus together with cisplatin, cetuximab and radiation in a phase I study. In patients judged by the medical oncologist as being unable to receive cisplatin, they will receive temsirolimus together with cetuximab and radiation in a separate arm in this phase I study. We will show the maximum tolerated doses of temsirolimus as a primary objective, with a secondary objective of examining progression-free survival at 12 months in each of these two arms.

ELIGIBILITY:
Inclusion Criteria:

Cohort A:

* Stage III or IVA-B HNC without prior RT except non-sm0kers with human papillomavirus (HPV) + nasopharynx and oropharynx. HPV+ oropharynx patients who have smoked regularly in the past 5 years are eligible.
* Patients with local or regional recurrence after surgery alone are eligible, as long as the recurrent stage is III or IVA-B
* Age > or = 18
* Karnofsky performance status > 70
* No severe active infection requiring intravenous antibiotics (oral antibiotics are allowable).
* Adequate renal function (creatinine < 1.5 mg/dl), based upon blood work performed within 1 month prior to registration.
* Adequate hepatic function (alkaline phosphatase and AST/ALT < 2 x ULN) based upon bloodwork performed within 1 month prior to registration.
* Adequate bone marrow function (ANC > 1.5; platelets > 100K) based upon blood work performed within one month prior to registration.
* Adequate cardiopulmonary function (no signs of acute coronary event and/or active CHF).
* No plans for other concurrent radiation therapy, chemotherapy or biologic anti-cancer therapy.

Cohort B:

* Platinum ineligible patients as defined by the multidisciplinary team.
* Stage III or IVA-B HNC without prior RT except nonsmokers with HPV + nasopharynx and oropharynx. HPV+ oropharynx patients who have smoked regularly in the past 5 years are eligible.
* Patients with local or regional recurrence after surgery alone are eligible, as long as the recurrent stage is III or IVA-B
* Age > or = 18
* KPS > 70
* No severe active infection requiring intravenous antibiotics (oral antibiotics are allowable).
* Adequate hepatic function (alkaline phosphatase and AST/ALT < 2 x ULN) based upon bloodwork performed within 1 month prior to registration.
* Adequate bone marrow function (ANC > 1.5; platelets > 100K) based upon bloodwork performed within one month prior to registration.
* Adequate cardiopulmonary function (no signs of acute coronary event and/or active CHF).
* No plans for other concurrent radiation therapy, chemotherapy or biologic anti-cancer therapy.

Exclusion Criteria:

* Current, recent (within 4 weeks of enrollment in this study) or planned participation in an experimental drug study other than this one.
* KPS < 70%
* Expected survival < 6 months
* Early stage head and neck cancer as defined as T1N0 or T2N0 by AJCC 7th edition
* Poorly controlled blood pressure, defined as systolic bp > 150 and/or diastolic bp > 100 despite medication.
* Unstable angina.
* NY Heart Association (NYHA) Grade II or greater congestive heart failure.
* History of myocardial infarction or stroke within 6 months.
* Clinically significant peripheral vascular disease.
* Evidence of bleeding diathesis or coagulopathy.
* Presence of brain or spinal cord metastases.
* Major surgical procedure(s), open biopsy or significant traumatic injury within 14 days prior to initiation of radiation therapy and/or anticipation of need for major surgical procedure during the course of the study.
* Minor surgical procedures such as needle/core biopsies, dental work, PEG placement, tracheostomy within 10 days prior to initiation of radiation therapy.
* Carotid artery exposure or other signs of impending carotid artery hemorrhage.
* History of abdominal fistula and/or gastrointestinal abdominal abscess within 6 months prior to enrollment.
* Serious, non-healing wound, ulcer, or bone fracture.
* Prior irradiation that would result in radiotherapy field "overlap."
* Requirement for high dose oral anticoagulation (i.e., goal INR > 2.0). "Mini-dose" anticoagulation may be used to assist in patency of central venous lines. Subcutaneous low-molecular weight heparin is allowable.
* No known allergies to any of the drug therapies being used in this protocol.
* No pregnancy, lactation or inability to use medically acceptable birth control if of childbearing potential.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-12-08 (Actual); Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Torisel | 7 weeks
  To determine the maximum tolerated dose (MTD) and a recommended phase II dose (RP2D) of Torisel (Torisel) when given with chemoradiotherapy (radiosensitized radiotherapy with cetuximab, cisplatin or both).

SECONDARY OUTCOMES:
Progression-Free Survival | 12 months
  Progression-free survival (PFS) rate at 12 months (PFS12)

CONTACTS AND LOCATIONS:
Overall Officials: Voichita Bar-Ad, MD, Principal Investigator — Thomas Jefferson University

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org